CLINICAL TRIAL: NCT03222401
Title: IGHID 11705 A Randomized, Open-label, Controlled Clinical Trial to Assess the Efficacy of F598 in Preventing an Experimental Urethral Infection With Neisseria Gonorrhoeae in Healthy Male Subjects
Brief Title: Trial to Assess the Efficacy of F598 in Preventing an Experimental Urethral Infection With N. Gonorrhoeae in Healthy Males
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis suggested that the trial, as designed, was not adequately powered to detect a therapeutic effect.
Sponsor: Alopexx Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Organization: AlopexxPharma (Unknown)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: AP-GC-201-16
Record Dates: First submitted 2017-07-07; First posted 2017-07-19 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Neisseria Gonorrhoeae

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled in 6 identical cohorts of 4 subjects each. Within each cohort, subjects will be randomized to:
  1. Control (n=1)
  2. F598, 1 mg/kg (n=1)
  3. F598, 3 mg/kg (n=1)
  4. F598, 10 mg/kg (n=1)
Who Masked: Participant
Masking Description: All doses of F598 will be administered on an open-label basis. Investigators will be unblinded, and subjects will be aware if they are randomized to the control group or one of the active dose groups; however, subjects in one of the active dose groups will not be informed of their randomized dosage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Control subjects will not receive an infusion or placebo
- 1 mg/kg single infusion of F598 (Experimental): 1 mg/kg single infusion of F598
  Interventions: Drug: 1 mg/kg single infusion of F598
- 3 mg/kg single infusion of F598 (Experimental): 3 mg/kg single infusion of F598
  Interventions: Drug: 3 mg/kg single infusion of F598
- 10 mg/kg single infusion of F598 (Experimental): 10 mg/kg single infusion of F598
  Interventions: Drug: 10 mg/kg single infusion of F598

INTERVENTIONS:
Drug: 1 mg/kg single infusion of F598 — 1 mg/kg single infusion of F598
  Other Names: F598
  Arms: 1 mg/kg single infusion of F598
Drug: 3 mg/kg single infusion of F598 — 3 mg/kg single infusion of F598
  Other Names: F598
  Arms: 3 mg/kg single infusion of F598
Drug: 10 mg/kg single infusion of F598 — 10 mg/kg single infusion of F598
  Other Names: F598
  Arms: 10 mg/kg single infusion of F598

SUMMARY:
Approximately 24 healthy male volunteers between the ages of 18 and 35 years will be enrolled at a single center for a duration of two months for each subject. Subjects who meet the enrollment criteria will be randomized to one of four open-label groups: Control (no treatment) or treatment with F598 at one of three doses. Following F598 administration or assignment to the Control group, subjects must return to the study site for inoculation with N. gonorrhoeae within 2 weeks. Once subjects have been inoculated with N. gonorrhoeae, they will enter the observation phase and will return to the study site daily for up to 5 days. At the end of the observation phase, definitive antibiotic therapy will be administered. A follow-up visit will be conducted 3-5 days after definitive antibiotic and a confirmatory interaction will occur with the subjects 7-10 days after the follow-up to confirm the subject's response. A final visit will occur approximately 8 weeks after inoculation.

DETAILED DESCRIPTION:
The study is comprised of 8 phases:

1. Screening (Visits 1 and 2)
2. F598 administration (Visit 3)
3. Inoculation (Visit 4)
4. Observation (Visits 5 - 8, as needed)
5. Definitive antibiotic treatment (Visit 9)
6. Test of cure (Visit 10)
7. Confirmatory interaction (Visit 11)
8. Final pharmacokinetic (PK)/pharmacodynamic (PD)/anti-drug antibody determination (Visit 12)

For the purposes of standardization, Day 1 of the study will be considered the day of inoculation.

During the Screening phase, prospective subjects will undergo informed consent and will be reviewed for their compatibility with the eligibility criteria. Those subjects who meet all of the Inclusion criteria and none of the Exclusion criteria will be enrolled. Following enrollment, subjects must undergo a repeat urine screen for C. trachomatis, N. gonorrhoeae and T. vaginalis (Days -17 to -4).

If the second urine screening test is negative, subjects will enter the F598 administration phase. Subjects will return to the study site and will be randomized to one of four open-label groups: Control (no treatment) or treatment with F598 at one of three doses. Following F598 administration or assignment to the Control group, subjects must return to the study site for inoculation with N. gonorrhoeae within 2 weeks. Thus, F598 will be administered on any one of Days -12 to -2.

During the inoculation phase, subjects will return to the study site and receive an inoculum of N. gonorrhoeae in the anterior urethra. A third and final urine screen for C. trachomatis, N. gonorrhoeae and T. vaginalis will be obtained immediately before inoculation.

Once subjects have been inoculated with N. gonorrhoeae, they will enter the observation phase and will return to the study site daily for up to 5 days for a physical examination (in particular, for evidence of urethral discharge) and a urine sample for evidence of infection (NAAT and culture) as well as blood for F598 PK/PD and safety labs.

The observation phase will end and definitive antibiotic therapy will be administered when any one of four criteria is met:

1. The subject requests antibiotic treatment
2. The subject is found to by symptomatic (discharge, urethral discomfort)
3. The subject has reached Day 6 of the study

Thus, depending on the circumstances, definitive antibiotic therapy can be administered between Days 2 - 6, inclusive.

A follow-up visit at the study site will be conducted 3 - 5 days after definitive antibiotic therapy has been administered to ensure treatment response. Thus, depending on when the subject received antibiotics, this visit could occur between Days 5 - 11, inclusive. A physical examination will be performed and urine for evidence of infection (NAAT) as well as blood for F598 PK/PD will be obtained.

A confirmatory interaction with the subject will occur at the study site 7 - 10 days after the follow-up visit to confirm the subject's response and answer any questions the subject may have. Thus, depending on when the subject had his follow-up visit, the confirmatory visit could occur between Days 12 - 21, inclusive. Blood for F598 PK/PD, anti-F598 antibodies and safety labs will be obtained.

A final visit will occur approximately 8 weeks after inoculation (days 52 - 60) to obtain serum for PK/PD and anti-F598 antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male between the ages of 18 and 35 years
2. Able and willing to be located easily by providing street address and telephone number (land line and/or cell phone number)
3. Able and willing to provide written informed consent
4. Able and willing to attend all study visits and follow-up visit during the week after treatment
5. Willing to abstain from masturbation during the 6 days after inoculation
6. Willing to abstain from all sexual activity during the course of the study
7. No clinically significant abnormalities on physical examination
8. No clinically significant abnormalities in serum chemistries, hematology and urinalysis
9. Urine negative for chlamydia, gonorrhea and trichomonas
10. No history of sexually transmitted infections (STIs), including syphilis and hepatitis B (HBV) & hepatitis C (HCV)
11. Negative human immunodeficiency virus (HIV), syphilis and HCV serologies
12. Negative HBV core and surface antibodies or results consistent with immunization (negative HBV core antibody/positive HBV surface antibody)
13. No history of bleeding diathesis
14. No history of seizures (due to reports of seizures with ciprofloxacin)
15. No history of cancer, except basal cell carcinoma of the skin more than 5 years ago
16. No history of drug abuse
17. No history of psychiatric disorders, except depression controlled by medication
18. No history of genitourinary surgery

Exclusion Criteria:

1. Student or employee under the direct supervision of any of the study investigators
2. Any known immunodeficiencies including complement deficiency, antibody deficiency, chronic granulomatous disease or HIV infection
3. Sickle cell disease
4. Psychiatric disorders that would interfere with the ability of the subject to comply with the requirements of the protocol
5. Unstable depression (defined as receiving either <3 months of the same medication (and dose) or a decompensating event during the previous 3 months) or depression that, in the opinion of the investigator, will compromise the subject's ability to comply with protocol requirements
6. Heart murmur or heart disease
7. Anatomic abnormality of the urinary tract
8. Any antibiotic treatment in the past 30 days, or azithromycin in the past 60 days
9. Chemotherapy within the past year
10. Current steroid use, except for topical application
11. Allergy to penicillin, cephalosporins, ciprofloxacin or to lidocaine
12. Treatment with medications that are contraindicated with cefixime, ceftriaxone or ciprofloxacin and that cannot be withheld for the single doses given in this study.

    1. Medications not permitted with cefixime or ceftriaxone include:

       * Warfarin
       * Probenecid
       * Aspirin
       * Diuretics such as furosemide
       * Aminoglycoside antibiotics
       * Chloramphenicol
    2. Medications not permitted with ciprofloxacin include:

       * Tizanidine
       * Theophylline
       * Warfarin
       * Glyburide
       * Cyclosporine
       * Probenecid
       * Phenytoin
       * Methotrexate
       * Antacids, multivitamins, and other dietary supplements containing magnesium, calcium, aluminum, iron or zinc
       * Caffeine-containing medications
       * Sucralfate or didanosine chewable or buffered
13. Major organ dysfunction
14. Any significant pre-existing condition preventing full compliance with the study
15. Infection or any serious underlying medical condition that would impair the ability of the subject to receive protocol treatment

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male between the ages of 18 and 35 years
Enrollment: 10 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of F598 in preventing an experimental urethral infection with N. gonorrhoeae | Through study completion, an average of two months
  Following the inoculation of N. gonorrhoeae, assess efficacy based of the proportion of infected subjects in each treatment group

SECONDARY OUTCOMES:
Assess the impact of F598 on urethritis symptoms caused by N. gonorrhoeae infection | Up to 6 weeks
  Urethritis signs as measured on targeted physical examination or symptoms reported by subject
Incidence of Treatment-Emergent Adverse Events [Safety and Immunogenicity] | Through study completion, an average of two months
  Monitor the treatment-emergent adverse events, infusion-associated reactions and anti-drug antibodies following administration of F598
Pharmacokinetic evaluation by measuring change from baseline in the concentration of F598 in the blood | Through study completion, an average of two months
  Cmax: Observed maximum serum concentration
Pharmacokinetic evaluation by measuring change from baseline in the concentration of F598 in the blood | Through study completion, an average of two months
  Tmax: Time to attain maximum serum concentration
Pharmacokinetic evaluation by measuring change from baseline in the concentration of F598 in the blood | Through study completion, an average of two months
  T 1/2: Elimination half-life
Pharmacokinetic evaluation by measuring change from baseline in the concentration of F598 in the blood | Through study completion, an average of two months
  AUC: Area under the serum concentration-time curve
Pharmacokinetic evaluation by measuring change from baseline in the concentration of F598 in the blood | Through study completion, an average of two months
  CL: Total body clearance of F598 from plasma
Pharmacokinetic evaluation by measuring change from baseline in the concentration of F598 in the blood | Through study completion, an average of two months
  V: Volume of F598 distribution at steady state
Pharmacodynamics: Associations between the PD parameters and infection rate | Through study completion, an average of two months
  Blood samples for serum bactericidal activity following administration of F598
Pharmacodynamics: Associations between the PD parameters and infection rate | Through study completion, an average of two months
  Blood samples for complement fixation following administration of F598

CONTACTS AND LOCATIONS:
Overall Officials: Hal Landy, MD, Study Director — Alopexx Pharmaceuticals, LLC
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No